CLINICAL TRIAL: NCT02309450
Title: Pilot Study to Assess Efficacy and Safety of a Triple Therapy With Asunaprevir, Daclatasvir and BMS-791325 in HCV Genotype 4-infected Patients After Failure of Pegylated Interferon-Ribavirin Regimen
Brief Title: Pilot Study to Assess Efficacy and Safety of a Triple Therapy With Asunaprevir, Daclatasvir, and BMS-791325 in HCV Genotype 4-infected Patients After Failure of Pegylated Interferon-Ribavirin Regimen
Acronym: QUATTROTURBO
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: BMS decision
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRSHC33QUATTROTURBO; 2014-002724-27 (EudraCT Number)
Record Dates: First submitted 2014-10-31; First posted 2014-12-05 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis C Virus Genotype 4 Infection
MeSH Terms: interventions — asunaprevir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Asunaprevir, Daclatasvir and BMS - 791325 (Experimental)
  Interventions: Drug: .Asunaprevir, Daclatasvir and BMS - 791325

INTERVENTIONS:
Drug: .Asunaprevir, Daclatasvir and BMS - 791325 — All patients will receive an all-oral HCV tritherapy with Asunaprevir (200mg), Daclatasvir (30mg) and BMS-791325 (75mg) in a fixed-dose combination (FDC) tablet, twice a day (1 tablet in the morning and 1 tablet in the evening) for 12 weeks.

SUMMARY:
ANRS HC 33 is a pilot study to assess efficacy and safety of a DCV 3DAA therapy with Asunaprevir, Daclatasvir and BMS-791325 in HCV genotype 4-infected patients after failure of pegylated Interferon-Ribavirin regimen.

Proportion of patients with cirrhosis will be limited to 50% of all patients included, cirrhosis being defined as a METAVIR score of F4 on the liver biopsy or an hepatic impulse elastometry ≥ 14 kPa or a Fibrotest® result > 0,75.

DETAILED DESCRIPTION:
The clinical trial is multi-centre, national, Phase 2, open-label, single-arm. The primary objective of this study is to assess, in HCV genotype 4-infected patients in failure to prior treatment with pegylated Interferon and Ribavirin bitherapy, the rate of sustained virological response (SVR) 12 weeks after 12 weeks of treatment with an all-oral combination of 3 DAAs in a Fixed-Dose-Combination (Asunaprevir 200 mg, Daclatasvir 30 mg and BMS - 791325 75 mg) twice a day.

Estimated enrollment is 60 patients during the enrolment period (9 months).

Schedule of assessments:

w4-w8 : screening D0 : Start of anti-HCV tritherapy (Asunaprevir + Daclatasvir + BMS-791325) w12: stop tritherapy w24: Sustained virological response SVR12 assessment (12 weeks post treatment) w36 : Sustained virological response SVR24 assessment (24 weeks post treatment)

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years
* Infection with HCV genotype 4, confirmed by detectable HCV RNA ≥ 1000 IU/ml at pre-inclusion
* Failure to a prior treatment with pegylated Interferon and Ribavirin, with failure being defined as follows:

  * Non-response: HCV viral load remaining detectable during and at the end of P/R treatment.
  * Relapse: undetectable HCV viral load during P/R treatment and detectable after the end of the treatment.
  * HCV breakthrough: undetectable HCV viral load during P/R treatment becoming detectable before the end of treatment.
* Anti-HCV treatment discontinued for at least the last 3 months
* Fibrosis at any stage, with documentation of the presence or absence of cirrhosis at the pre-inclusion visit:

  * history of liver biopsy showing cirrhosis lesions (METAVIR F4), at any time in the patient's history, or
  * good quality (length ≥ 1 cm and ≥ 5 portal spaces) liver biopsy dating from less than 18 months to establish the METAVIR, or
  * hepatic impulse elastometry (Fibroscan®) dating from less than 6 months and of good quality (at least 10 measurements on an incidence with IQR of less than 30% of the median elastometry measured and a success rate of 60%) or
  * interpretable Fibrotest® dating from less than 6 months The proportion of patients with cirrhosis will be limited to 50% of all patients included, cirrhosis being defined as a METAVIR score of F4 on the liver biopsy or an hepatic impulse elastometry ≥ 14 kPa or a Fibrotest® result > 0,75.
* Men and women of a child-bearing age and their heterosexual partners must use adequate contraception during treatment and up to 8 weeks after the end of treatment for women, 12 weeks after the end of treatment for men.
* Written informed consent signed by the patient and the investigator (on the day of the pre-inclusion at the latest and before any examination required by the study) (article L1122-1-1 Public Health Code)
* Patients with Health insurance (Sécurité Sociale or Couverture Médicale Universelle)

Exclusion Criteria:

Medical history

* CHILD B or C cirrhosis
* Previous HCV therapy including HCV NS3 protease inhibitor, and/or HCV NS5A replication complex inhibitor and/or HCV NS5B polymerase inhibitor

Current condition

* Positive HBs Antigen
* Confirmed HIV-1 or HIV-2 infection
* Pregnant or breast-feeding women
* Transplant recipients
* Any evolutive ongoing malignant disease, including hepatocellular carcinoma, which will be specifically screened for before inclusion
* Consumption of alcohol which, in the investigator's opinion, will be an obstacle to the patient's participation and to his/her remaining in the study
* Drug addiction which, in the investigator's opinion, will be an obstacle to the patient's participation and to his/her remaining in the study. Patients included in a programme of substitution with methadone or buprenorphine could be included. The opinion of an addictology consultant is recommended for patients presenting with current drug use or drug use in the past year.
* Patients taking part in another clinical trial during the 30 days prior to inclusion
* Patient under guardianship, trusteeship or judicial protection

Biological criteria

* ALT ≥ 5xULN
* Total bilirubin ≥ 34 µmol/L, unless a documented history of Gilbert's disease
* Hb < 85 g/L
* Platelets < 50 000/mm3
* Kidney failure defined by creatinine clearance < 50mL/mn (MDRD formula)
* QTc > 440 msec for males or 460 msec for females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
HCV sustained virological response rate | week 24
  The primary endpoint is the Sustained Virological Response Rate defined by an undetectable HCV RNA at W24, that is to say 12 weeks after the end of the DCV 3DAA therapy associating Asunaprevir, Daclatasvir and BMS - 791325 (SVR12). In case of premature total or partial interruption of HCV treatment, the primary endpoint will also be assessed at week 24.

SECONDARY OUTCOMES:
Number of patients with adverse events | up to week 36
Treatment interruptions | from day 0 to week12
  Number of patients who totally or partially interrupt,treatment
Causes of treatment discontinuation | form day 0 to week 12
  toxicity or side effects
Self-reported symptoms | Day 0, week 12, week 36
  self-questionnaire (ANRS AC24 perceived symptoms scale)
Patients adherence rate | week 4, week 12
  measured using the (ANRS) self -questionnaire
HCV viral load | day 0, week 1, week 2, week 4, week 8, week 12, week 16, week 20, week 24, week 36.
Evaluation of the relationship between HCV subtypic distribution at baseline (by sequencing of the HCV NS5B domain) and the virological kinetics and response | at screening
Proportion of patients with resistance mutations to Asunaprevir and/or Daclatasvir and/or BMS in case of virological failure | up to week 12
Child-Pugh score (composite measure) | at screening
  For cirrhotic patients
  Encephalopathy None+1 Mild to moderate (grade 1 or 2)+2 Severe (grade 3 or 4)+3
  Ascites None+1 Mild to moderate (diuretic responsive)+2 Severe (diuretic refractory)+3
  Bilirubin (mg/dL) < 2+1 2-3+2 > 3+3
  Albumin (g/dL) > 3.5+1 2.8-3.5+2 < 2.8+3
  International normalized ratio < 1.7+1 1.7-2.3+2 > 2.3+3 Total score of 5-6 = Grade A (well compensated disease) Total score of 7-9 = Grade B (disease with significant functional compromise) Total score of 10-15 = Grade C (decompensated liver disease)
Insulin resistance measured using the HOMA-IR score | Day 0, week 36
Parameters that define metabolic syndrome | Day 0, week 36
Evolution of liver fibrosis | Day 0, week 36
  Fibrotest® or imaging Fibroscan®. Fibrosis will be evaluated with the same method (Fibroscan® or Fibrotest®) at baseline and week 36.
MELD score (composite measure) | at screening
  For cirrhotic patients
  MELDScore = 10 * ((0.957 * ln(Creatinine)) + (0.378 * ln(Bilirubin)) + (1.12 * ln(INR))) + 6.43

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Roulot, MD, Principal Investigator — Hopital Avicenne, APHP
Locations (1):
- France, All the Regions of the Country, France